CLINICAL TRIAL: NCT02429622
Title: A Phase Ⅰ/Ⅱ Study of Simultaneous Integrated Boost Radiotherapy and Concurrent Chemotherapy in Patients With Locally Advanced Esophageal Carcinoma
Brief Title: Simultaneous Integrated Boost Radiotherapy and Concurrent Chemotherapy for Locally Advanced Esophageal Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zefen Xiao, Professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-133/923
Record Dates: First submitted 2015-04-24; First posted 2015-04-29 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Esophageal Neoplasms
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Paclitaxel; nedaplatin; Esophagectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Radical 2.14 (Experimental): Radiation：Patients undergo radiotherapy once daily 5 days a week for an average of 5.5 weeks in the absence of disease progression or unacceptable toxicity. IMRT simultaneous integrated boost technique is used to achieve a prophylactic dosage and radical dosage of 1.8Gy and 2.14Gy once respectively.
  Concurrent chemotherapy:Patients may receive a dosage range of Paclitaxel from 45 to 60 mg/m2 and Nedaplatin 25mg/m2 per week in the following 5 weeks after enrollment with radiotherapy at the same time in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: IMRT simultaneous integrated boost; Drug: Paclitaxel; Drug: Nedaplatin
- Radical 2.17 (Experimental): Radiation：Patients undergo radiotherapy once daily 5 days a week for an average of 5.5 weeks in the absence of disease progression or unacceptable toxicity. IMRT simultaneous integrated boost technique is used to achieve a prophylactic dosage and radical dosage of 1.8Gy and 2.17Gy once respectively.
  Concurrent chemotherapy:Patients may receive a dosage range of Paclitaxel from 45 to 60 mg/m2 and Nedaplatin 25mg/m2 per week in the following 5 weeks after enrollment with radiotherapy at the same time in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: IMRT simultaneous integrated boost; Drug: Paclitaxel; Drug: Nedaplatin
- Radical 2.21 (Experimental): Radiation：Patients undergo radiotherapy once daily 5 days a week for an average of 5.5 weeks in the absence of disease progression or unacceptable toxicity. IMRT simultaneous integrated boost technique is used to achieve a prophylactic dosage and radical dosage of 1.8Gy and 2.21Gy once respectively.
  Concurrent chemotherapy:Patients may receive a dosage range of Paclitaxel from 45 to 60 mg/m2 and Nedaplatin 25mg/m2 per week in the following 5 weeks after enrollment with radiotherapy at the same time in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: IMRT simultaneous integrated boost; Drug: Paclitaxel; Drug: Nedaplatin
- Neoadjuvant 2.14 (Experimental): Radiation：Patients undergo radiotherapy once daily 5 days a week for an average of 4.5 weeks in the absence of disease progression or unacceptable toxicity. IMRT simultaneous integrated boost technique is used to achieve a prophylactic dosage and radical dosage of 1.8Gy and 2.14Gy once respectively.
  Concurrent chemotherapy:Patients may receive a dosage range of Paclitaxel from 45 to 60 mg/m2 and Nedaplatin 25mg/m2 per week in the following 4 weeks after enrollment with radiotherapy at the same time in the absence of disease progression or unacceptable toxicity. Assessment of surgery: Patients eligible for surgery after multiple disciplinary consultation will receive esophagectomy after a 4-6 weeks break after chemoradiation in the absence of any contraindication.
  Interventions: Radiation: IMRT simultaneous integrated boost; Drug: Paclitaxel; Drug: Nedaplatin; Procedure: Esophagectomy

INTERVENTIONS:
Radiation: IMRT simultaneous integrated boost — To achieve a prophylactic dosage and radical dosage once respectively
Drug: Paclitaxel — Paclitaxel from 45 to 60 mg/m2 per week concurrent with radiotherapy for 5weeks
  Other Names: Taxel
Drug: Nedaplatin — Nedaplatin 25mg/m2 per week concurrent with radiotherapy for 5weeks
Procedure: Esophagectomy — Radical esophagectomy 4-6 weeks after neoadjuvant therapy
  Arms: Neoadjuvant 2.14

SUMMARY:
This phase Ⅰ/Ⅱ trial is designed to explore a higher radiation dose by using IMRT simultaneous integrated boost technique with or without concurrent chemotherapy for locally advanced esophageal carcinoma.

DETAILED DESCRIPTION:
Despite the application of IMRT and the studies of concurrent chemoradiation in esophageal carcinoma, which improves 5-year survival rate from 10% to 20%-40% and decrease recurrence rate from 80% to 50%-60%, local recurrence remains to be the most common failure pattern. Therefore, enhancing local control is the key to obtain a better survival.

A phase Ⅱ study of radical radiotherapy with IMRT simultaneous integrated boost technique and concurrent chemotherapy for esophageal carcinoma use the same radiation dose as the high dose arm in RTOG 94-05, which reveals an significantly improved median survival time of 23 months and 3-year overall survival rate of 44.4%. This study implies the simultaneous integrated boost technique may be effective to some extent. But the question is how to identify patients who may gain potential benefits, and whether this therapeutic model can be copied in the specific situation in China? Few adverse effects such as perforation, hemorrhage and stenosis was reported, mainly owing to the lack of cases. For widely application of this new technique in the clinic, more studies need to be conducted in the future to obtain sufficient evidence.

The current IMRT can simultaneously achieve prophylactic dose (DT 50Gy) and radical dose (DT 60-64Gy) in respective target volume by using inverse intensity-modulated planning system. However, it is still controversial on whether esophageal carcinoma can receive prescription dose more than 2.0Gy each time. That is to say, it is challengeable to find an optimal fraction dose and total dose between tumor and adverse effects. For this reason, the dose escalation trial is to be conducted to explore the clinical value and optimal dose to esophageal carcinoma with different radiosensitivity, and also provide data support for phase Ⅲ clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of clinical stage T2-4N0-1M1a untreated squamous esophageal carcinoma
* KPS≥70
* Adequate organ function
* No known history of drug allergy

Exclusion Criteria:

* Known drug allergy
* Insufficient hepatorenal function
* Severe cardiovascular diseases, diabetes with uncontrolled blood sugar, mental disorders, uncontrolled severe infection, active ulceration which need intervention.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-01; Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | up to 3 years

SECONDARY OUTCOMES:
Overall survival (OS) | up to 5 years

OTHER OUTCOMES:
Adverse events | up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Zefen Xiao, MD, Principal Investigator — The Department of Radiation Oncology ,Cancer Institute & Hospital，Chinese Academy of Medical Science
Locations (1):
- Zefen Xiao, Beijing, Beijing Municipality, China

REFERENCES:
- [Result] Cooper JS, Guo MD, Herskovic A, Macdonald JS, Martenson JA Jr, Al-Sarraf M, Byhardt R, Russell AH, Beitler JJ, Spencer S, Asbell SO, Graham MV, Leichman LL. Chemoradiotherapy of locally advanced esophageal cancer: long-term follow-up of a prospective randomized trial (RTOG 85-01). Radiation Therapy Oncology Group. JAMA. 1999 May 5;281(17):1623-7. doi: 10.1001/jama.281.17.1623. PMID 10235156
- [Result] Welsh J, Settle SH, Amini A, Xiao L, Suzuki A, Hayashi Y, Hofstetter W, Komaki R, Liao Z, Ajani JA. Failure patterns in patients with esophageal cancer treated with definitive chemoradiation. Cancer. 2012 May 15;118(10):2632-40. doi: 10.1002/cncr.26586. Epub 2011 Oct 5. PMID 22565611
- [Result] Minsky BD, Pajak TF, Ginsberg RJ, Pisansky TM, Martenson J, Komaki R, Okawara G, Rosenthal SA, Kelsen DP. INT 0123 (Radiation Therapy Oncology Group 94-05) phase III trial of combined-modality therapy for esophageal cancer: high-dose versus standard-dose radiation therapy. J Clin Oncol. 2002 Mar 1;20(5):1167-74. doi: 10.1200/JCO.2002.20.5.1167. PMID 11870157
- [Result] Yu WW, Zhu ZF, Fu XL, Zhao KL, Mao JF, Wu KL, Yang HJ, Fan M, Zhao S, Welsh J. Simultaneous integrated boost intensity-modulated radiotherapy in esophageal carcinoma: early results of a phase II study. Strahlenther Onkol. 2014 Oct;190(11):979-86. doi: 10.1007/s00066-014-0636-y. Epub 2014 Mar 8. PMID 24609941
- [Derived] Li C, Ni W, Wang X, Zhou Z, Deng W, Chang X, Chen D, Feng Q, Liang J, Wang X, Deng L, Wang W, Bi N, Zhang T, Xiao Z. A phase I/II radiation dose escalation trial using simultaneous integrated boost technique with elective nodal irradiation and concurrent chemotherapy for unresectable esophageal Cancer. Radiat Oncol. 2019 Mar 15;14(1):48. doi: 10.1186/s13014-019-1249-5. PMID 30876442